CLINICAL TRIAL: NCT02635698
Title: Opti-WIN: Effectiveness of the Optifast Program Compared With a Reduced-energy Food Based Diet Plan on Body Weight
Brief Title: Effectiveness of the Optifast Program Compared With a Reduced-energy Food Based Diet Plan on Body Weight
Acronym: Opti-WIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14.21.CLI
Record Dates: First submitted 2015-12-11; First posted 2015-12-21 (Estimated); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group, Optifast (Experimental): OPTIFAST, medically supervised weight-management program
  Interventions: Other: Optifast
- Control group, Low-energy, low-fat (Active Comparator): Food-based program, current standard of care for weight management
  Interventions: Other: Food-Based

INTERVENTIONS:
Other: Optifast — medically-supervised weight management program
  Arms: Intervention group, Optifast
Other: Food-Based — low-energy, low-fat diet
  Arms: Control group, Low-energy, low-fat

SUMMARY:
Compare percent change in loss of body weight between the OPTIFAST program and a food-based energy-deficit program

ELIGIBILITY:
Inclusion Criteria:

* Adult males and females between 18 and 70 years
* Obese (BMI > 30 kg/m2 and 55 kg/m2)
* Non-smokers or smoking cessation > 6 months
* < 14 alcoholic beverages per week
* Willing and able to give informed consent

Exclusion Criteria:

* Active participation in any weight loss program within previous 3 months
* Weight changes of > 5% body weight within previous 3 months
* Participated in an Optifast program within prior 5 years
* Prior bariatric surgery or liposuction
* Use of any medication prescribed for weight loss in the past 3 months
* Current major disease or GI disease that is poorly controlled (Crohn's, ulcerative colitis)
* Type 1 DM
* Current ESRD
* Current COPD
* Any major or active hepatic disease requiring inpatient or outpatient treatment
* History of acute pancreatitis in the past year
* Active cancer treatment in the past 2 years other than non-malignant skin cancers
* Uncontrolled hypertension (Blood pressure 160/100 or greater)
* Hemoglobin A1c > 10%
* Recent CV event in past 6 months
* Pregnancy, childbirth, or nursing within prior 6 months
* Eating Attitudes Test (EAT-26) > 30
* Current major depressive disorder with Center for Epidemiological Studies Depression Scale-Revised (CESD-R) score > 16
* Schizophrenia, history of bipolar disorder
* Recent hospitalization for psychiatric illness in past 6 months
* Dependence on alcohol or sedative-hypnotic drugs
* Intolerance or allergy to Optifast product
* Unable to read/speak English
* Orthopedic limitation preventing participation in regular physical activity
* Untreated thyroid disease, abnormal TSH, non on stable dose of hormone replacement for hyperthyroidism
* Major surgery defined as any surgical procedure that might require prolonged convalescence or limit participation in the program in any way
* Inability to complete the 7-day run-in satisfactorily

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2015-11; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Percent weight change | 26 weeks
  Percent change in body weight between Initial Visit/Baseline and 26 weeks
Percent weight change | 52 weeks
  Percent change in body weight between Initial Visit/Baseline and 52 weeks

SECONDARY OUTCOMES:
Ability to meet weight goals | 52 weeks
  Percentage of subjects meeting short- and long-term weight loss goals
Change in anthropometrics | 52 weeks
  change in BMI in kg/m^2 from baseline to 52 weeks
Change in cardiometabolic outcomes | 52 weeks
  Change in 10-year cardiovascular risk score (% likelihood to develop CVD in 10 years)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Alaska Premier Health, Anchorage, Alaska
  - Alexian Brothers Weight Loss Solutions, Schaumburg, Illinois
  - University of Michigan Health System, Ann Arbor, Michigan
  - Brody School of Medicine, East Carolina University, Greenville, North Carolina
  - Wake Forest School of Medicine, Winston-Salem, North Carolina
  - Neuro-Behavioral Clinical Research, Inc., Canton, Ohio
  - Central Ohio Nutrition Center, Inc., Gahanna, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Houston Center for Clinical Research, Sugar Land, Texas

REFERENCES:
- [Derived] Ard JD, Lewis KH, Rothberg A, Auriemma A, Coburn SL, Cohen SS, Loper J, Matarese L, Pories WJ, Periman S. Effectiveness of a Total Meal Replacement Program (OPTIFAST Program) on Weight Loss: Results from the OPTIWIN Study. Obesity (Silver Spring). 2019 Jan;27(1):22-29. doi: 10.1002/oby.22303. Epub 2018 Nov 13. PMID 30421863